CLINICAL TRIAL: NCT06299020
Title: Risks of Intermittent Fasting in Patients With Primary Adrenal Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital La Rabta (Other)
Responsible Party: Principal Investigator, Melika Chihaoui, professor, Hopital La Rabta
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HLaRabta24
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Primary Adrenal Insufficiency; Intermittent Fasting
Keywords: continuous glucose monitoring; Hypoglycemia; Dehydration
MeSH Terms: conditions — Addison Disease; Intermittent Fasting; Hypoglycemia; Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non fasting (No Intervention): Non fasting arm: usual diet and behavior
- Fasting (Experimental): Intermittent fasting
  Interventions: Behavioral: intermittent fasting

INTERVENTIONS:
Behavioral: intermittent fasting — fasting from predawn to sunset (no eating and no drinking), for approximately 16 hours.
  Other Names: Ramadan fasting
  Arms: Fasting

SUMMARY:
In primary adrenal insufficiency, there is an increased risk of hypoglycaemia and dehydration. These risks have been little studied particularly during intermittent fasting. The present study aimed to assess these risks in a prospective study of 30 subjects with primary adrenal insufficiency. Patients will undergo a clinical examination, blood sampling and continuous glucose monitoring for fourteen days (one week of fasting and one week of non-fasting).

DETAILED DESCRIPTION:
The risk of hypoglycaemia in primary adrenal insufficiency (PAI) is well known but has been only few studied. It is explained by cortisol insufficiency. Only a few publications concerned this subject. The risk of hypoglycaemia seems to be increased during acute decompensation, following cessation of treatment and during fasting or delayed food intake. So, this risk would be increased during intermittent fasting such as the Ramadan fast. A previous study carried out in the endocrinology department of La Rabta University Hospital involving 30 subjects with secondary adrenal insufficiency who were monitored by continuous glucose monitoring (CGM) for 24 hours showed three cases of hypoglycaemia during intermittent fasting and no hypoglycaemia outside fasting. Studies assessing the risks of intermittent fasting concerned subjects with secondary adrenal insufficiency. No study assessed the risks of intermittent fasting in PAI. Furthermore, given the mineralocorticoid deficiency in PAI, there is also a risk of dehydration and hypotension.

Aims of the study:

Overall objective: to assess the risks of intermittent fasting in subjects with primary adrenal insufficiency.

Specific objectives:

* To assess the frequency of hypoglycaemia in subjects with primary adrenal insufficiency during fasting and outside fasting.
* To assess the frequency of dehydration in subjects with primary adrenal insufficiency during fasting and outside fasting.
* To study the factors associated with hypoglycaemia and dehydration.

Methods :

Type of study: prospective, cross over, comparative study with subjects taken as their own controls.

A group of 15 patients will be studied during the week preceding the month of Ramadan (non fasting week) and the first week of Ramadan (fasting week). A group of 15 patients will be studied during the fourth week of Ramadan (fasting week) and the first week after Ramadan (non fasting week). The analysis will thus concern 210 fasted days and 210 non-fasted days.

The included patients will be examined on two occasions 14 days apart. Visit 1 will include a clinical examination, the setting up of the continuous glucose monitoring system, a fasting blood sampling and the delivery of monitoring sheets.

Clinical data:

* Demographic data: age, gender
* Data relating to PAI: age, aetiology, replacement therapy. Fasting history and course (number of days fasted, occurrence of complications).
* Quality of life and quality of sleep questionnaire.
* weight, height, waist circumference, supine and standing blood pressure, heart rate, presence of melanoderma, signs of dehydration.

The patient will be given dietary and hygiene advice on fasting and the treatment (gluco- and mineral-corticosteroids) will be adjusted if necessary, in accordance with the recommendations published in 2021 and 2022.

Biological data: urea, iono

During the study period (two weeks), patients will be asked to fill in a monitoring form which will include details of medication taken, waking and bedtimes, physical activity and the occurrence of any discomfort (asthenia, signs of hypoglycaemia, signs of arterial hypotension or other).

Patients will be monitored during the fasting period by one of the investigators by telephone in order to check compliance with the protocol and the possible occurrence of complications.

Criteria for breaking the fasting: occurrence of malaise during fasting, hypoglycaemia diagnosed by CGM, elevation of urea or hyperkalaemia.

Visit 2 : the patients will undergo a clinical examination including quality of life and quality of sleep questionnaires and a physical examination, fasting blood sampling, recovery of the continuous glucose monitoring system and monitoring sheets.

Diagnosis criteria:

* Hypoglycaemia is defined as interstitial glucose measured during CGM < 2.8mmol/l.
* Dehydration is defined by the presence of arterial hypotension (BP <9/6cmHg or orthostatic hypotension) or elevated plasma urea.

ELIGIBILITY:
Inclusion Criteria:

* Primary adrenal insufficiency
* Disease duration of at least one year
* Substituted with hydrocortisone and fludrocortisone
* Wishing to fast during the month of Ramadan 2024

Exclusion Criteria:

* Diabetes mellitus
* Renal insufficiency
* Hepatic insufficiency
* Cardiac insufficiency
* Respiratory insufficiency
* Use of hypoglycaemic agents
* Use of diuretics
* Use of glucocorticoids other than those prescribed for replacement
* Poor control of the disease (asthenia, malaise, melanoderma, discontinuation of treatment, etc.)
* Pregnancy
* Breast-feeding.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
hypoglycemia | the fasting period from predawn to sunset (approximately 16 hours)
  clinical signs or interstitial glucose lower than 2.8mmol/l

SECONDARY OUTCOMES:
Dehydration | the fasting period from predawn to sunset (approximately 16 hours)
  clinical signs of dehydration or increase of plasmatic urea

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital La Rabta, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after the publication
Access Criteria: by mail

REFERENCES:
- [Result] Lee SC, Baranowski ES, Sakremath R, Saraff V, Mohamed Z. Hypoglycaemia in adrenal insufficiency. Front Endocrinol (Lausanne). 2023 Nov 20;14:1198519. doi: 10.3389/fendo.2023.1198519. eCollection 2023. PMID 38053731
- [Result] Kawahara T, Tsuji M, Tominaga N, Toyama N, Toda M. Frequency of Adrenal Insufficiency in Patients With Hypoglycemia in an Emergency Department: A Cross-sectional Study. J Endocr Soc. 2022 Aug 4;6(10):bvac119. doi: 10.1210/jendso/bvac119. eCollection 2022 Oct 1. PMID 36042975
- [Result] Watanabe T, Ozawa A, Ishii S, Tomaru T, Shibusawa N, Saito T, Yamada E, Horiguchi K, Nakajima Y, Matsumoto S, Yoshino S, Katano-Toki A, Hashimoto K, Mori M, Okada S, Satoh T, Yamada M. Usage of continuous glucose monitoring (CGM) for detecting an unrecognized hypoglycemia and management of glucocorticoid replacement therapy in adult patients with central hypoadrenalism. Endocr J. 2018 May 28;65(5):547-556. doi: 10.1507/endocrj.EJ16-0387. Epub 2018 Apr 4. PMID 29618670
- [Result] Chihaoui M, Grira W, Bettaieb J, Yazidi M, Chaker F, Rejeb O, Oueslati I, Feki M, Kaabachi N, Slimane H. The risk for hypoglycemia during Ramadan fasting in patients with adrenal insufficiency. Nutrition. 2018 Jan;45:99-103. doi: 10.1016/j.nut.2017.07.014. Epub 2017 Aug 3. PMID 29129244
- [Result] Chihaoui M, Yazidi M, Oueslati I, Khessairi N, Chaker F. Intermittent fasting in adrenal insufficiency patients: a review and guidelines for practice. Endocrine. 2021 Oct;74(1):11-19. doi: 10.1007/s12020-021-02804-z. Epub 2021 Jul 2. PMID 34213700
- [Result] Hussain S, Hussain S, Mohammed R, Meeran K, Ghouri N. Fasting with adrenal insufficiency: Practical guidance for healthcare professionals managing patients on steroids during Ramadan. Clin Endocrinol (Oxf). 2020 Aug;93(2):87-96. doi: 10.1111/cen.14250. Epub 2020 Jun 15. PMID 32419166
- [Derived] Chihaoui M, Sta J, Kamoun E, Belhadjsliman C, Khessairi N, Oueslati I, Yazidi M, Chaker F, Feki M. Hypoglycaemia and other risks of ramadan fasting in patients with primary adrenal insufficiency: A prospective controlled trial using 24-hour glucose monitoring. J Endocrinol Invest. 2025 Oct 18. doi: 10.1007/s40618-025-02728-9. Online ahead of print. PMID 41108503